CLINICAL TRIAL: NCT00939250
Title: A Comprehensive Intervention for Diabetes and Comorbid Depression in Primary Care
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Madhukar H. Trivedi, MD, Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STU 042009-010; R34DK081031 (NIH)
Record Dates: First submitted 2009-07-13; First posted 2009-07-14 (Estimated); Last update posted 2020-09-02 (Actual); Status verified 2020-09

CONDITIONS: Type 2 Diabetes; Major Depressive Disorder
Keywords: Diabetes; Depression; Disease Self Management; Measurement Based Care
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Depressive Disorder, Major; Diabetes Mellitus; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Diabetes and depression intervention (Experimental): Measurement based care for diabetes and depression, disease self management for diabetes and depression
  Interventions: Behavioral: Diabetes and depression intervention
- Diabetes intervention (Active Comparator): Measurement based care for diabetes, disease self management for diabetes
  Interventions: Behavioral: Diabetes intervention

INTERVENTIONS:
Behavioral: Diabetes and depression intervention — Disease self management for diabetes and depression
  Other Names: Measurement based care; Disease self management
  Arms: Diabetes and depression intervention
Behavioral: Diabetes intervention — Disease self management for diabetes
  Other Names: Measurement based care; Disease self management
  Arms: Diabetes intervention

SUMMARY:
The study involves a 32-week randomized controlled trial in primary care of a comprehensive diabetic and depression intervention in patients with type 2 diabetes and comorbid MDD, compared to a group treated with usual care for MDD plus disease self-management and measurement-based care for diabetes.

DETAILED DESCRIPTION:
The overarching goal of the study is to translate research-based treatment procedures that have been shown to improve outcomes for both DM and MDD for use in primary care. More specifically, the aims are: 1) to evaluate the benefits of CDDI in improving diabetic outcomes compared to usual care for MDD plus disease self-management for diabetes; 2) to evaluate the benefits of CDDI in improving depression outcomes compared to the UC for MDD treatment protocol; and 3) to evaluate the benefits of CDDI in terms of improved (1) cardiovascular risk factors (blood pressure, body mass index, lipids, and abdominal fat), (2) levels of exercise and better diet, (3) clinician and patient satisfaction with care, (4) fidelity to treatment guidelines, and (5) cognitive function.

ELIGIBILITY:
Inclusion Criteria:

* Meets DSM-IV criteria for single or recurrent nonpsychotic MDD, and whom the physician deems it necessary to start on an antidepressant.
* Meets clinical criteria for type 2 diabetes as follows: (1) on pharmacological treatment for type 2 diabetes and/or (2) fasting plasma glucose > 126mg/dL on 2 separate occasions or an abnormal oral glucose tolerance test (OGTT) (2-hours post load glucose ≥ 200mg/dL).
* HbA1C > 7
* Ability and willingness to provide written informed consent
* Hamilton Rating Scale for Depression (HRSD) score ≥ 14
* Not on antidepressant medication for at least 2 weeks prior to screen (or 6 weeks in the case of fluoxetine or monoamine oxidase inhibitors - MAOIs)

Exclusion Criteria:

* Women who are pregnant or breastfeeding
* Type 1 diabetes
* General medical conditions that contraindicate use of antidepressant medications
* Unstable medical illnesses, such as uncontrolled hypertension or symptomatic cardiovascular disease, such as congestive heart failure or angina
* Current or past psychotic disorders including bipolar disorder (I, II, or NOS), schizophrenia, or schizoaffective disorder; anorexia; bulimia
* High risk for being unable to complete the study due to hospitalization, suicide attempts, significant self-mutilation, or other self-injurious or destructive behavior
* Concomitant pharmacological or psychotherapeutic treatment including but not limited to anxiolytics, neuroleptics, mood stabilizers, and/or other agents without proven antidepressant efficacy; cognitive behavioral therapy; current use of other medications that would be contraindicated with antidepressant treatment, as determined by the study doctor
* History of current substance or alcohol dependence requiring detoxification within the last 6 months
* Currently suicidal or considered a high suicide risk
* Require inpatient treatment for their depression

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-10; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Glycosylated Hemoglobin | week 16, 32

SECONDARY OUTCOMES:
Quick Inventory of Depressive Symptoms - Self Report | week 16, 32

CONTACTS AND LOCATIONS:
Overall Officials: Madhukar H. Trivedi, M.D., Principal Investigator — University of Texas Southwestern Medical Center; David W. Morris, Ph.D., Study Director — University of Texas Southwestern Medical Center
Locations (1):
- Family and Community Medicine Clinic, University of Texas Southwestern Medical Center, Dallas, Texas, United States